CLINICAL TRIAL: NCT02053337
Title: A Randomised Cross-over Clinical Evaluation to Compare Performance of ALLEVYN◊ Life and Mepilex™ Border Dressings on Patient Well-being Related Endpoints.
Brief Title: A RCT to Compare Performance of Two Foam Dressings on Patient Well-being Related Endpoints.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CE047ALF
Record Dates: First submitted 2014-01-20; First posted 2014-02-03 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self adhesive foam dressing (Experimental): Sponsor manufactured self adhesive foam dressing. Use of CE marked dressing according to instructions for use and study protocol.
  Interventions: Device: Self adhesive foam dressing
- Comparator self adhesive foam dressing (Active Comparator): Non Sponsor manufactured self adhesive foam dressing. Use of CE marked dressing according to instructions for use and study protocol.
  Interventions: Device: Self adhesive foam dressing

INTERVENTIONS:
Device: Self adhesive foam dressing — Self adhesive foam dressing
  Other Names: ALLEVYN◊ Life

SUMMARY:
ALLEVYN◊ Life and Mepilex™ Border are both layered foam dressings with a silicone adhesive wound contact layer. Both are indicated for the same uses; however ALLEVYN◊ Life has a number of attributes designed to meet a range of characteristics associated with principles of wellbeing.

The aim for this evaluation is to assess, in a clinical setting and against a number of identified criteria, the performance of the ALLEVYN◊ Life dressing compared to Mepilex™ Border in terms of characteristics of the attributes of wellbeing.

◊ Trademark of Smith & Nephew

™ All trademarks acknowledged

ELIGIBILITY:
Inclusion Criteria:

Patients ≥18 years old

Males and females (females must not be pregnant and must use contraception if of child bearing potential.)

Presence of a single suitable wound which can be the reference wound without treatment impacting on any other wound(s) on the patient.

Presence of a suitable wound which can be treated with the available sizes and shapes of ALLEVYN◊ Life (10.3cm X 10.3cm, 12.9cm X 12.9cm, 15.4cm X 15.4cm, 21cm X 21cm) and Mepilex™ Border (7cm X 7.5cm, 10cm X 12.5cm, 15cm X 17.5, 17cm X 20cm)

Presence of an exuding wound of at least 6 weeks duration at the point of enrolment, healing by secondary intention

The patient is able to understand the evaluation and is willing to consent to the evaluation.

The patient is available to participate for the anticipated duration of the evaluation.

Exclusion Criteria:

Patients with confirmed or suspected clinically infected reference wounds.

Patients with wounds that, in the opinion of the clinician, is likely to heal within a time period of 4 weeks from point of enrolment.

Patients with a reference wound undergoing treatment with compression therapy.

Patients where a reference wound cannot be treated in isolation from other wounds.

Patients with deep reference wounds that, in the opinion of the clinician, necessitate filler material.

Patients with a known sensitivity to any of the constituents of the evaluation products.

Patients with a known history of poor compliance with medical treatment.

Patients who have participated in this evaluation previously and have been withdrawn from the study.

Patients unable to understand or speak the English language.

Patients without the capacity to understand and answer wellbeing related questions

Females who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Subjective rating of the impact of the dressing performance and characteristics on patient wellbeing (referred to as patient wellbeing score) | After (up to) 10 days of dressing wear
  The primary outcome, a subjective patient wellbeing/preference score, is calculated using a combination of responses from 8 individual questions on a patient questionnaire and 2 further dressing retention related measures at the end of treatment with each dressing (up to maximum of 10 days). Individual patient questions relate to the effect of specific dressing performance /characteristics on patient wellbeing (each on a 0-10 scale: 0 = most negative response, 10 = most positive response).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ousey, Principal Investigator — University of Huddersfield
Locations (1):
- Northumbria NHS, Newcastle, United Kingdom